CLINICAL TRIAL: NCT00129714
Title: A Randomized Controlled Trial of Conservative Therapy in Cervical Radiculopathy
Brief Title: Westeinde Brachialgia Study
Acronym: WEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Center Haaglanden (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 542
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Radiculopathy, Cervical
Keywords: cervical radiculopathy conservative treatment
MeSH Terms: conditions — Radiculopathy | interventions — Physical Therapy Modalities

ARMS (3):
- wait and see (No Intervention)
- collar (Experimental)
  Interventions: Other: cervical collar
- physiotherapy (Experimental)
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: cervical collar
  Arms: collar
Other: physiotherapy
  Arms: physiotherapy

SUMMARY:
The Westeinde Brachialgia Study (WEB) is a randomized controlled trial to establish the effect of cervical collar or physiotherapy compared to a wait-and-see policy in patients with acute cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical radiculopathy caused by spondylosis or disc protrusion is a common disorder with a usually benign natural course. Often, physiotherapy (exercise programs) and/or cervical collar are prescribed. However, there are no reliable data on the effects of these conservative therapies.

In this study, patients with acute cervical radiculopathy, defined by clinical criteria, are randomized for cervical collar, physiotherapy or a wait-and-see policy.

ELIGIBILITY:
Inclusion Criteria:

* Cervical radiculopathy defined by neck pain irradiating to one arm with at least one of the following: provocation by neck movements or sensory changes in one or more adjacent dermatomes or diminished deep tendon reflexes in the affected arm; or muscle weakness in one or more adjacent myotomes.

Exclusion Criteria:

* Arm pain existing longer than one month
* Clinical signs of spinal cord compression
* Previously treated with physiotherapy or a cervical collar

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2003-08; Primary Completion 2007-04 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
pain and disability at 3 and 6 weeks and at 6 months

SECONDARY OUTCOMES:
time back to work
persistent signs and symptoms
surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jos TJ Tans, MD PhD, Study Chair — Medical Center Haaglanden
Locations (3):
- Netherlands (3):
  - Meander Medical Center, Amersfoort
  - Groene Hart Ziekenhuis, Gouda
  - Medical Center Haaglanden, The Hague

REFERENCES:
- [Derived] Kuijper B, Tans JT, Beelen A, Nollet F, de Visser M. Cervical collar or physiotherapy versus wait and see policy for recent onset cervical radiculopathy: randomised trial. BMJ. 2009 Oct 7;339:b3883. doi: 10.1136/bmj.b3883. PMID 19812130
- [Derived] Kuijper B, Tans JT, Schimsheimer RJ, van der Kallen BF, Beelen A, Nollet F, de Visser M. Degenerative cervical radiculopathy: diagnosis and conservative treatment. A review. Eur J Neurol. 2009 Jan;16(1):15-20. doi: 10.1111/j.1468-1331.2008.02365.x. PMID 19087147